CLINICAL TRIAL: NCT04129476
Title: Effect of a Cooperative Education Program Based on Precede-Proceed Model During Pregnancy on Postpartum Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gonabad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Atefeh Dehnoalian, Principal Investigator, Gonabad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GonabadUMS
Record Dates: First submitted 2019-10-09; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Post Partum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooperative Education Program (Experimental): We explore the effects of a cooperative education program based on precede-proceed model during pregnancy on preventing postpartum depression.
  Interventions: Behavioral: Cooperative Education Program based on Precede-Proceed Model
- Control (No Intervention): We provide routine care for these people during pregnancy

INTERVENTIONS:
Behavioral: Cooperative Education Program based on Precede-Proceed Model — The study population is pregnant women in Gonabad city between 30 and 35 weeks of gestation. In the experimental group, the training program was based on the PRECEDE-PROCEDURE model, including training on anatomy and prenatal physiology, prenatal and postnatal care, prenatal and postnatal mental health, as well as prenatal and postnatal events, and Mothers' feelings and attitudes, as well as postpartum problems and strategies will be discussed. The training period is 60 minutes in 4 consecutive sessions. Predisposing, reinforcing and enabling factors inventory, General health questionnaire (GHQ), Edinburgh depression inventory Will be filled Before the intervention, immediately after the intervention and 4 to 6 weeks after the intervention.
  Arms: Cooperative Education Program

SUMMARY:
This trail aims to evaluate the effects of a cooperative education program based on precede-proceed model during pregnancy on preventing postpartum depression in southern Razavi Khorasan Province.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate in the research
* Gestational age 30-35 weeks
* Be literate
* No history of depression or mental illness in the past
* Healthy fetus on ultrasound

Exclusion Criteria:

* Having a preterm birth
* Refusal to attend training sessions

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum Depression | Edinburgh Postnatal Depression Scale will be filled from baseline to 6 week
  Depression in POSTPARTUM WOMEN, usually within four weeks after giving birth (PARTURITION). The degree of depression ranges from mild transient depression to neurotic or psychotic depressive disorders. It includes 10 questions and each question is scored from 0 to 3. The total score ranges from 0 to 30 and a score of 10-13 indicates mild postpartum depression while a score of 14-15 indicates moderate postpartum depression. Score of 16 or higher is considered as severe depression which necessitates introduction to a psychologist.

SECONDARY OUTCOMES:
Predisposing, reinforcing and enabling factors inventory | Before the intervention, immediately after the intervention and 4 to 6 weeks after the intervention.
  for this section, a questionnaire was designed based on a literature review and according to educational and ecological Phase of precede-proceed model. Predisposing factors will be measured using 10 and 18 questions regarding knowledge and attitude, respectively. The second section of the questionnaire will be related to the enabling factors which were measured through 6 questions. Yes or no questions were designed and scored as follows: no=1, somewhat=2, yes=3. The third section of the questionnaire measures reinforcing factors through 2 questions with yes, no and somewhat answers being scored as 2, 0 and 1, respectively.
General health questionnaire (GHQ) | Before the intervention, immediately after the intervention and 4 to 6 weeks after the intervention.
  The General Health Questionnaire (GHQ) is a screening device for identifying minor psychiatric disorders in the general population and within community or non-psychiatric clinical settings such as primary care or general medical out-patients.it consists of 4 subscales including physical symptoms, anxiety symptoms, social functioning and depressive symptoms. Each scale is made of 7 questions which are assessed based on a Likert scale scoring as never (0), few (1), high (2) and very high (3). The total score for each person ranges from 0 to 84. Cutoff point for the questionnaire is reported to be 23. In this method, individuals with score of 23 or less are considered healthy and those with score of 24 or higher are suspected to be mentally disordered.

CONTACTS AND LOCATIONS:
Overall Officials: Baloochi, Study Chair — Gonabad University of Medical Science
Locations (1):
- Gonabad University of Medical Science, Gonābād, Khorasan Razavi, Iran

IPD SHARING:
Plan to Share IPD: No